CLINICAL TRIAL: NCT00819091
Title: A Randomized, Double-blind, Placebo-controlled Parallel Group Efficacy and Safety Study of BI 1356 (5 mg Administered Orally Once Daily) Over 18 Weeks in Type 2 Diabetic Patients With Insufficient Glycaemic Control (HbA1c 7.0-10%) Despite Background Therapy With a Sulfonylurea Drug.
Brief Title: Randomized, Double-blind (db), Placebo-controlled 18 Week Study of Linagliptin (BI 1356) in Type 2 Diabetic Patients With Insufficient Glycaemic Control on a Sulfonylurea Drug
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.35; 2008-003118-86 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2011-08-01 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- BI 1356 (Active Comparator): 5 mg orally (po) once daily
  Interventions: Drug: BI 1356
- Placebo (Placebo Comparator): one tablet once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1356 — 5mg orally (po) tablet qd
  Arms: BI 1356
Drug: Placebo — Placebo matching BI 1356 5mg one tablet daily
  Arms: Placebo

SUMMARY:
Efficacy and safety of BI 1356 compared to placebo in patients with type 2 diabetes who have insufficient glycaemic control despite treatment with a sulfonylurea drug.

ELIGIBILITY:
Inclusion criteria:

Patients between 18 and 80 years old with type 2 diabetes and insufficient glycemic control [glycosylated hemoglobin (HbA1c 7% to 10%)] despite therapy with a sulfonylurea drug

Exclusion criteria:

Myocardial infarction,stroke or transient ischaemic attack in last 6 months Treatment with rosiglitazone, pioglitazone, GLP-1 analogues, insulin or anti-obesity drugs in the past 3 months Impaired hepatic function Severe renal impairment Current treatment with systemic steroids Change in thyroid hormone dosage Hereditary galactose intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (45):
- United States (13):
  - 1218.35.10002 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1218.35.10001 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1218.35.10016 Boehringer Ingelheim Investigational Site, National City, California
  - 1218.35.10017 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1218.35.10021 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1218.35.10013 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1218.35.10015 Boehringer Ingelheim Investigational Site, Flint, Michigan
  - 1218.35.10018 Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - 1218.35.10004 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1218.35.10005 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1218.35.10020 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1218.35.10009 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.35.10019 Boehringer Ingelheim Investigational Site, Sugar Land, Texas
- Argentina (4):
  - 1218.35.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1218.35.54005 Boehringer Ingelheim Investigational Site, Corrientes
  - 1218.35.54001 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 1218.35.54006 Boehringer Ingelheim Investigational Site, Parque Velez Sarfield
- Hungary (5):
  - 1218.35.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.35.36002 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.35.36004 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.35.36005 Boehringer Ingelheim Investigational Site, Budapest
  - 1218.35.36003 Boehringer Ingelheim Investigational Site, Debrecen
- India (8):
  - 1218.35.91003 Boehringer Ingelheim Investigational Site, Aligarh, Uttar Pradesh
  - 1218.35.91007 Boehringer Ingelheim Investigational Site, Aminjikarai, Tamilnadu
  - 1218.35.91001 Boehringer Ingelheim Investigational Site, Bangalore, Karnataka
  - 1218.35.91004 Boehringer Ingelheim Investigational Site, Bangalore, Karnataka
  - 1218.35.91002 Boehringer Ingelheim Investigational Site, Indore
  - 1218.35.91008 Boehringer Ingelheim Investigational Site, Mumbai, Maharastra
  - 1218.35.91005 Boehringer Ingelheim Investigational Site, Nagpur, Maharashtra
  - 1218.35.91006 Boehringer Ingelheim Investigational Site, Pune, Maharastra
- Japan (3):
  - 1218.35.81003 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.35.81001 Boehringer Ingelheim Investigational Site, Shinjyuku-ku,Tokyo
  - 1218.35.81002 Boehringer Ingelheim Investigational Site, Suita, Osaka,
- Poland (5):
  - 1218.35.48002 Boehringer Ingelheim Investigational Site, Bialystok
  - 1218.35.48004 Boehringer Ingelheim Investigational Site, Lublin
  - 1218.35.48003 Boehringer Ingelheim Investigational Site, Poznan
  - 1218.35.48001 Boehringer Ingelheim Investigational Site, Rzeszów
  - 1218.35.48005 Boehringer Ingelheim Investigational Site, Wroclaw
- Russia (7):
  - 1218.35.70008 Boehringer Ingelheim Investigational Site, Arkhangelsk
  - 1218.35.70001 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.35.70002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.35.70003 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.35.70006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.35.70009 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1218.35.70007 Boehringer Ingelheim Investigational Site, Yaroslavl

REFERENCES:
- [Derived] McGill JB, Barnett AH, Lewin AJ, Patel S, Neubacher D, von Eynatten M, Woerle HJ. Linagliptin added to sulphonylurea in uncontrolled type 2 diabetes patients with moderate-to-severe renal impairment. Diab Vasc Dis Res. 2014 Jan;11(1):34-40. doi: 10.1177/1479164113507068. Epub 2013 Oct 29. PMID 24169807
- [Derived] Lewin AJ, Arvay L, Liu D, Patel S, von Eynatten M, Woerle HJ. Efficacy and tolerability of linagliptin added to a sulfonylurea regimen in patients with inadequately controlled type 2 diabetes mellitus: an 18-week, multicenter, randomized, double-blind, placebo-controlled trial. Clin Ther. 2012 Sep;34(9):1909-19.e15. doi: 10.1016/j.clinthera.2012.07.008. Epub 2012 Aug 29. PMID 22939034
- [Derived] Johansen OE, Neubacher D, von Eynatten M, Patel S, Woerle HJ. Cardiovascular safety with linagliptin in patients with type 2 diabetes mellitus: a pre-specified, prospective, and adjudicated meta-analysis of a phase 3 programme. Cardiovasc Diabetol. 2012 Jan 10;11:3. doi: 10.1186/1475-2840-11-3. PMID 22234149

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo tablet taken orally once daily
- Linagliptin (BI 1356) 5.0 mg: Linagliptin 5.0 mg tablet taken orally once daily
Period: Overall Study
Arm/Group | Placebo | Linagliptin (BI 1356) 5.0 mg
Started | 84 | 161
Completed | 77 | 151
Not Completed | 7 | 10
Not completed — Adverse Event | 3 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Linagliptin 5.0 mg: Linagliptin 5.0 mg tablet taken orally once daily
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 5.0 mg | Total
Number analyzed (Participants) | 84 | 161 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.2) | 57.2 (9.8) | 56.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 84 | 116
  Male | 52 | 77 | 129
Race/Ethnicity, Customized [Number; unit: participants]
  White | 34 | 73 | 107
  Black | 6 | 11 | 17
  Asian | 43 | 76 | 119
  American Indian/Alaskan Native | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic | 70 | 133 | 203
  Hispanic | 14 | 28 | 42
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/square meter] | 28.21 (5.12) | 28.40 (5.02) | 28.33 (5.04)
Baseline glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage] | 8.6 (0.72) | 8.61 (0.85) | 8.61 (0.81)
Fasting blood plasma glucose (FPG) [Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)] | 174.9 (49.0) | 182.0 (51.8) | 179.6 (50.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) at Week 18
Description: HbA1c is measured as a percent. The change from baseline reflects the Week 18 HbA1c percent minus the Week 0 HbA1c percent. Means are adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline, week 18
Population: Full Analysis Set includes all randomized patients with baseline and on-treatment value of HbA1c. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 82 | 158
percent | -0.07 (0.10) | -0.54 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model includes treatment and number of prior oral anti-diabetic drug as fixed classification effects and baseline HbA1c as a linear covariate; Least Squares Mean Difference = -0.47, 95% CI [-0.70 to -0.24], Standard Error of Mean 0.12

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 18
Description: Change from baseline reflects the Week 18 FPG minus the Week 0 FPG. Means are adjusted for baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline, week 18
Population: Full Analysis Set includes all randomized patients with baseline and on-treatment value of FPG. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 78 | 155
mg/dL | -1.8 (4.5) | -8.2 (3.3)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.2406, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -6.4, 95% CI [-17.2 to 4.3], Standard Error of Mean 5.5

3. Secondary Outcome: Percentage of Patients With Absolute Efficacy Response (HbA1c < 7%) at Week 18
Description: An absolute efficacy response is defined as HbA1c < 7.0% at 18 weeks. A non-response is defined as HbA1c >= 7.0% at 18 weeks.
Time Frame: week 18
Population: FAS patients with baseline HbA1c >= 7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: Percentage of Patients
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 82 | 158
Percentage of Patients
  HbA1c < 7% | 3.7 | 15.2
  HbA1c >= 7% | 96.3 | 84.8
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.0065, Regression, Logistic; Odds Ratio (OR) = 6.466, 95% CI [1.684 to 24.825]

4. Secondary Outcome: Percentage of Patients With Absolute Efficacy Response (HbA1c < 6.5%) at Week 18
Description: An absolute efficacy response is defined as HbA1c < 6.5% at 18 weeks. A non-response is defined as HbA1c >= 6.5% at 18 weeks.
Time Frame: week 18
Population: FAS patients with baseline HbA1c >= 6.5%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 82 | 158
percentage of participants
  HbA1c < 6.5% | 2.4 | 5.7
  HbA1c >= 6.5% | 97.6 | 94.3
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.2431, Regression, Logistic; Odds Ratio (OR) = 2.653, 95% CI [0.515 to 13.652]

5. Secondary Outcome: Percentage of Patients With HbA1c Lowering by at Least 0.5% From Baseline at Week 18
Description: An efficacy response is defined as HbA1c lowered by 0.5% or more at 18 weeks. A non-response is defined as HbA1c not lowered by 0.5% or more at 18 weeks.
Time Frame: Baseline, week 18
Population: FAS patients. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 82 | 158
percentage of participants
  HbA1c lower by at least 0.5% | 22 | 57.6
  HbA1c not lower by at least 0.5% | 78.0 | 42.4
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.125, 95% CI [2.747 to 9.562]

6. Secondary Outcome: Mixed Model Repeated Measurements Analysis of Change From Baseline in HbA1c at Week 6
Description: HbA1c is measured as a percent. The change from baseline reflects the Week 6 HbA1c percent minus the Week 0 HbA1c percent. Means are adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline, week 6
Population: FAS patients. Mixed Model Repeated Measurements (MMRM) analysis of Observed Cases (OC).
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 82 | 158
percent | -0.02 (0.07) | -0.43 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM with treatment, number oral anti-diabetic drugs, week within patients, week-treatment interaction and baseline HbA1c as a linear covariate; Least Squares Mean Difference = -0.41, 95% CI [-0.585 to -0.230]

7. Secondary Outcome: Mixed Model Repeated Measurements Analysis of Change From Baseline in HbA1c at Week 12
Description: HbA1c is measured as a percent. The change from baseline reflects the Week 12 HbA1c percent minus the Week 0 HbA1c percent. Means are adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline, week 12
Population: FAS patients. Mixed Model Repeated Measurements (MMRM) analysis of Observed Cases (OC).
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 82 | 158
percent | -0.11 (0.09) | -0.61 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.50, 95% CI [-0.720 to -0.276]

8. Secondary Outcome: Mixed Model Repeated Measurements Analysis of Change From Baseline in HbA1c at Week 18
Description: as for outcome 1
Time Frame: Baseline, week 18
Population: FAS patients. Mixed Model Repeated Measurements (MMRM) analysis of Observed Cases (OC).
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 82 | 158
percent | -0.08 (0.10) | -0.55 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Least Squares Mean Difference = -0.47, 95% CI [-0.716 to -0.226]

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 6
Description: Change from baseline reflects the Week 6 FPG minus the Week 0 FPG. Means are adjusted for baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline, week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 78 | 155
mg/dL | -7.6 (3.8) | -13.5 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.197, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -5.9, 95% CI [-14.9 to 3.1], Standard Error of Mean 4.6

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: Change from baseline reflects the Week 12 FPG minus the Week 0 FPG. Means are adjusted for baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline, week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5.0 mg
Number analyzed (Participants) | 78 | 155
mg/dL | 4.1 (4.7) | -10.3 (3.4)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5.0 mg; Linagliptin 5.0 mg versus placebo; Test type: Superiority or Other; p = 0.0105, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -14.5, 95% CI [-25.5 to -3.4], Standard Error of Mean 5.6

ADVERSE EVENTS:
Time Frame: From day of first dose until 7 days after last dose
Arm/Group | Placebo | Linagliptin 5.0 mg
Serious Adverse Events (participants affected / at risk) | 1/84 | 5/161
Other Adverse Events (participants affected / at risk) | 14/84 | 14/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=84) | Linagliptin 5.0 mg (N=161)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=84) | Linagliptin 5.0 mg (N=161)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.